CLINICAL TRIAL: NCT05229055
Title: Intranasal Ketamine Versus Subcutaneous Ketamine for Treatment of Post Traumatic Acute Pain in the Emergency Department
Brief Title: Intranasal Ketamine Versus Subcutaneous Ketamine for Treatment of Post-traumatic Acute Pain in the Emergency Department ( INVESCK )
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Monastir Emergency departement, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Intranasal ketamine
Record Dates: First submitted 2021-11-20; First posted 2022-02-08 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: The intranasal route Ketamine solution was used. Applying a nasal spray pump where each spray delivered 20 mg of ketamine. After initial evaluation, each patient having the inclusion criteria receives one pulverisation (0.4 ml) per nostril of ketamine corresponding to a total dose of 20 mg of ketamine.
  The subcutaneous route :
  Ketamine dosing by subcutanous route was based on previous reports use for post operative pain management. . The results of these reports revealed that low-dose ketamine 20-60 mg (0.5mg/kg for patients weighing 40-120 kg) showed an over all decrease in either the amount of opioid used or the amount of pain experienced (10, 11). For our study, we decided to chose a dose of 20mg of ketamine for all patients administered via 1ml insulin syringe once subcutaneously.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: After initial medical evaluation, every patient who meet the inclusion criteria, will receive randomly either subcutaneous or intanasal dose of ketamine as detailed above according to the predetermined randomization. To ensure a double-blind administration of ketamine ; patients enrolled in the intranasal ketamine group will receive concomitantly 1ml of normal saline solution subcutaneously, and patients enrolled in the subcutaneous ketamine group will receive concomitantly a spray of normal saline solution in each nostril. None of the treating physician or nurses are aware about the medication received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal ketamine (Active Comparator): Ketamine solution 250 mg/5ml was used. It was applied intranasally using a nasal spray pump whereeach spray delivered approximately 0.4 ml of solution corresponding to 20 mg of ketamine. After initial evaluation, each patient having the inclusion criteria receives one pulverisation (0.4 ml) per nostril of ketamine corresponding to a total dose of 20 mg of ketamine. Ketamine dosing was based on previous reports of intranasal ketamine use in ED patients, doses ranged from 0.45mg/kg to 1.25mg/kg (9).
  Interventions: Drug: Ketamine
- subcutanous ketamine (Active Comparator): Ketamine dosing by subcutanous route was based on previous reports use for post operative pain management. . The results of these reports revealed that low-dose ketamine 20-60 mg (0.5mg/kg for patients weighing 40-120 kg) showed an over all decrease in either the amount of opioid used or the amount of pain experienced (10, 11).For our study, we decided to chose a dose of 20mg of ketamine for all patients administered via 1ml insulin syringe once subcutaneously.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — giving ketamine intranasal
  Other Names: ketalar

SUMMARY:
Pain is the most common complaint for emergency department (ED) visit. Intranasal ketamine has been shown to provide rapid, well-tolerated, effective analgesia to emergency department (ED) patients with acute pain. few trials have studied ketamine infusion subcutaneously for pain management in trauma patients.

DETAILED DESCRIPTION:
Materials and methods :

Study design It is a randomized, prospective, double blind, controlled, multicentric trial.

Study setting and selection of participants :

The trial is conducted in three community teaching hospitals :

* Emergency department, fattouma bourgiba university hospital, monastir, tunisia.
* Emergency department, sahloul university hospital, sousse, tunisia.
* Emergency department, farhat hached university hospital, sousse, tunisia.

Inculsion criteria :

The study includes patients aged 18 to 60 years who presented to the ED with acute limb trauma pain with a visual analgesic scale (VAS) of 5 or more on a standard 11 point (0-10). An informed consent is necessary. Pain was considered traumatic if it is reported as appearing immediately after the trauma and no anterior pain was described in the same limb.

The intranasal route Ketamine solution 250 mg/5ml was used. It was applied intranasally using a nasal spray pump where each spray delivered approximately 0.4 ml of solution corresponding to 20 mg of ketamine. After initial evaluation, each patient having the inclusion criteria receives one pulverisation (0.4 ml) per nostril of ketamine corresponding to a total dose of 20 mg of ketamine. Ketamine dosing was based on previous reports of intranasal ketamine use in ED patients, doses ranged from 0.45mg/kg to 1.25mg/kg.

The subcutaneous route :

Ketamine dosing by subcutanous route was based on previous reports use for post operative pain management. . The results of these reports revealed that low-dose ketamine 20-60 mg (0.5mg/kg for patients weighing 40-120 kg) showed an over all decrease in either the amount of opioid used or the amount of pain experienced. the investigators decided to chose a dose of 20mg of ketamine for all patients administered via 1ml insulin syringe once subcutaneously.

Protocol :

After initial medical evaluation, every patient who meet the inclusion criteria, will receive randomly either subcutaneous or intanasal dose of ketamine as detailed above according to the predetermined randomization. To ensure a double-blind administration of ketamine ; patients enrolled in the intranasal ketamine group will receive concomitantly 1ml of normal saline solution subcutaneously, and patients enrolled in the subcutaneous ketamine group will receive concomitantly a spray of normal saline solution in each nostril. None of the treating physician or nurses are aware about the medication received. The included patients were followed and monitored until their discharge from the ED. All enrolled patients underwent close supervision of study staff to ensure safety. Study investigators record VAS, and adverse effects at 15, 30, 60, 90, and 120 minutes and at ED discharge. During ED stay, patients were monitored in order to evaluate the need for rescue analgesic treatment. At 30 minutes, if patients report a pain numeric rating scale score of 5 or greater and request additional pain relief, titrated morphine is adminstered as a rescue analgesic with a dose of 0.1mg/kg repeated every 3 to 5 minutes if the pain numeric rating scale score is still greater or equal to 3.

. Patients's informed consent is obtained.

ELIGIBILITY:
Inclusion Criteria:

* • Patients who presented to the ED with acute limb trauma pain with a visual analgesic scale (VAS) of 5 or more on a standard 11 point (0-10).

  * Pain was considered traumatic if it is reported as appearing immediately after the trauma and no anterior pain was described in the same limb.

Exclusion Criteria:

* Pregnancy/Breastfeeding

  * altered mental status (GCS<15)
  * Allergy to ketamine or morphine
  * Weight less than 40 kg or greater than 100kg
  * Unstable vital signs (systolic blood pressure <90 or > 180mmHg, pulse rate<50 or >150bpm, and respiration rate <10 or >30 breath/min)
  * Medical history of acute head or eye injury
  * Medical history of seizure
  * Medical history of intracranial hypertension,
  * Medical history of chronic pain,
  * Medical history of severe renal or hepatic insufficiency.
  * Medical history of glaucoma
  * Alcohol or drug abuse
  * Psychiatric illness,
  * Recent (4 hours before) analgesic agent use.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
VAS decrease of more than 50% comparing to initial value at 30 minutes following analgesia administration | 30 minutes
  resolution of pain with decrease of VAS more than 50% comparing to initial value
rate of severe adverse events | 120 minutes
  occurence of severe adverse events

SECONDARY OUTCOMES:
rate of rescue analgesia 1 doses of morphine required to reach efficient analgesia | 30 minutes
  The need for rescue analgesia
rate of rescue analgesia 2 doses of morphine required to reach efficient analgesia | 120 minutes
  The need for rescue analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, Professor, Principal Investigator — University of Monastir
Locations (1):
- university of Monastir, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Todd KH, Ducharme J, Choiniere M, Crandall CS, Fosnocht DE, Homel P, Tanabe P; PEMI Study Group. Pain in the emergency department: results of the pain and emergency medicine initiative (PEMI) multicenter study. J Pain. 2007 Jun;8(6):460-6. doi: 10.1016/j.jpain.2006.12.005. Epub 2007 Feb 15. PMID 17306626
- [Background] Guirimand F, Dupont X, Brasseur L, Chauvin M, Bouhassira D. The effects of ketamine on the temporal summation (wind-up) of the R(III) nociceptive flexion reflex and pain in humans. Anesth Analg. 2000 Feb;90(2):408-14. doi: 10.1097/00000539-200002000-00031. PMID 10648330
- [Background] Schmid RL, Sandler AN, Katz J. Use and efficacy of low-dose ketamine in the management of acute postoperative pain: a review of current techniques and outcomes. Pain. 1999 Aug;82(2):111-125. doi: 10.1016/S0304-3959(99)00044-5. PMID 10467917
- [Background] Andolfatto G, Willman E, Joo D, Miller P, Wong WB, Koehn M, Dobson R, Angus E, Moadebi S. Intranasal ketamine for analgesia in the emergency department: a prospective observational series. Acad Emerg Med. 2013 Oct;20(10):1050-4. doi: 10.1111/acem.12229. PMID 24127709
- [Background] Galinski M, Dolveck F, Combes X, Limoges V, Smail N, Pommier V, Templier F, Catineau J, Lapostolle F, Adnet F. Management of severe acute pain in emergency settings: ketamine reduces morphine consumption. Am J Emerg Med. 2007 May;25(4):385-90. doi: 10.1016/j.ajem.2006.11.016. PMID 17499654
- [Background] Strigo IA, Duncan GH, Bushnell CM, Boivin M, Wainer I, Rodriguez Rosas EM, Persson J. The effects of racemic ketamine on painful stimulation of skin and viscera in human subjects. Pain. 2005 Feb;113(3):255-264. doi: 10.1016/j.pain.2004.10.023. PMID 15661431
- [Background] Smith DC, Mader TJ, Smithline HA. Low dose intravenous ketamine as an analgesic: a pilot study using an experimental model of acute pain. Am J Emerg Med. 2001 Oct;19(6):531-2. doi: 10.1053/ajem.2001.27152. No abstract available. PMID 11593484
- [Background] Andolfatto G, Innes K, Dick W, Jenneson S, Willman E, Stenstrom R, Zed PJ, Benoit G. Prehospital Analgesia With Intranasal Ketamine (PAIN-K): A Randomized Double-Blind Trial in Adults. Ann Emerg Med. 2019 Aug;74(2):241-250. doi: 10.1016/j.annemergmed.2019.01.048. Epub 2019 Mar 27. PMID 30926189
- [Background] Shrestha R, Pant S, Shrestha A, Batajoo KH, Thapa R, Vaidya S. Intranasal ketamine for the treatment of patients with acute pain in the emergency department. World J Emerg Med. 2016;7(1):19-24. doi: 10.5847/wjem.j.1920-8642.2016.01.003. PMID 27006733
- [Background] Tuchscherer J, McKay WP, Twagirumugabe T. Low-dose subcutaneous ketamine for postoperative pain management in Rwanda: a dose-finding study. Can J Anaesth. 2017 Sep;64(9):928-934. doi: 10.1007/s12630-017-0914-0. Epub 2017 Jun 19. PMID 28631150
- [Background] Elia N, Tramer MR. Ketamine and postoperative pain--a quantitative systematic review of randomised trials. Pain. 2005 Jan;113(1-2):61-70. doi: 10.1016/j.pain.2004.09.036. PMID 15621365